CLINICAL TRIAL: NCT04294290
Title: AN OPEN LABEL PHASE I STUDY OF hCT-MSC, AN UMBILICAL CORD-DERIVED MESENCHYMAL STROMAL CELL PRODUCT IN YOUNG CHILDREN WITH AUTISM SPECTRUM DISORDER
Brief Title: Open Label Phase I hCT-MSC in Toddlers With Autism Spectrum Disorder
Acronym: TACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Principal Investigator, Joanne Kurtzberg, MD, Jerome Harris Distinguished Professor of Pediatrics, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104460
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; ASD; Autism; PDD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hCT-MSC infusion (Experimental): hCT-MSC infusion
  Interventions: Biological: hCT-MSC infusion

INTERVENTIONS:
Biological: hCT-MSC infusion — This is a single site, phase I, open-label, prospective study of one intravenous infusion of human umbilical cord tissue-derived mesenchymal stromal cells (hCT-MSC) in 12 toddlers 18 to 48 months of age with autism spectrum disorder (ASD).

SUMMARY:
This is a single site, prospective study of one intravenous infusion of human umbilical cord tissue-derived mesenchymal stromal cells (hCT-MSC) in toddlers with autism spectrum disorder (ASD). Toddlers 18 to 48 months of age with a confirmed diagnosis of ASD will be eligible to participate. Diagnosis will be confirmed at the time of the eligibility visit at the Duke Center for Autism and Brain Development. All participants will receive a single intravenous dose of 2x106/kg hCT-MSC per kilogram at baseline. Assessments will be conducted at baseline and 6 months, with remote follow-up assessments at 12 months.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate safety and feasibility. Safety assessments include monitoring of acute infusion reactions, adverse events, incidence of infections, and markers of alloimmunization. Clinical outcome measures will also be described. A key clinical outcome measeure is the change in social communication abilities from baseline to 6 months based on the Joint Engagement Rating Inventory (JERI), a commonly-used and well-validated coding system for rating the quality and quantity of social communication skills in toddlers with and without ASD.91 JERI coding rates social communication abilities on a 1 to 7 scale and factors in both the quantity and quality of skills. The total joint engagement score as well as ratings on all JERI subscales that comprise the total score will be described.

Other clinical endpoints will include the PDD Behavior Inventory (PDDBI) autism composite score, the mean of the Socialization Subscale Standard Score and Communication Subscale Standard Score on the Vineland Adaptive Behavior Scales (VABS-3), the Clinical Global Impression Scale (CGI) - Severity and Improvement Scales, the Communicative Development Inventories (CDI-2): Words & Sentences subscales, attention abilities via eye-tracking, and brain activity.

Exploratory clinical endpoints will include autism symptoms measured by an app that elicits and records autism symptoms on an iPad (SenseToKnow), Autism Diagnostic Observation Scale (ADOS-2) Calibrated Severity Score (overall, social affect, and repetitive behavior), PDD Behavior Inventory (PDDBI) Subscales, and VABS-3 Standard Score and age equivalent for the following subscales: Socialization, Communication, and Daily Living and the Standard Score and age equivalent for the VABS-3 Adaptive Behavior Composite.

Safety and VABS-3 assessments will also be conducted remotely at three and 12 months. Duration of study participation will be 12 months from the time of the baseline infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 months to ≤ 48 months (48 months, 29 days) at the time of consent
2. Confirmed clinical DSM-5 diagnosis of Autism Spectrum Disorder using the DSM-5 Checklist as informed by the Autism Diagnostic Observation Schedule - 2.
3. Fragile X testing performed and negative; CMA and/or whole exome sequencing performed and results not linked to autism diagnosis
4. Stable on current psychoactive medication regimen (dose and dosing schedule) for at least 2 months prior to infusion of study product
5. Normal absolute lymphocyte count (≥1500/uL)
6. Participant and parent/guardian are English speaking
7. Able to travel to Duke University for two multi-day visits (baseline and six months) and parent/guardian is able to participate in interim surveys and interviews
8. Parental consent

Exclusion Criteria:

1. General:

   1. Review of medical records indicates ASD diagnosis not likely
   2. Screening data suggests that participant would not be able to comply with the requirements of the study procedures as assessed by the study team
   3. Family is unwilling or unable to commit to participation in all study-related assessments, including protocol follow up
   4. Sibling is enrolled in this (Duke hCT-MSC) study
2. Genetic:

   1. Records indicate that child has a known genetic syndrome such as (but not limited to) Fragile X syndrome, neurofibromatosis, Rett syndrome, tuberous sclerosis, PTEN mutation, cystic fibrosis, muscular dystrophy or a genetic mutation known to be associated with ASD
   2. Known pathogenic mutation or copy number variation (CNV) associated with ASD (e.g., 16p11.2, 15q13.2, 2q13.3)
3. Infectious:

   1. Known active CNS infection
   2. Evidence of uncontrolled infection based on records or clinical assessment
   3. Known HIV positivity
4. Medical:

   1. Known metabolic disorder
   2. Known mitochondrial dysfunction
   3. History of unstable epilepsy or uncontrolled seizure disorder, infantile spasms, Lennox Gastaut syndrome, Dravet syndrome, or other similar chronic seizure disorder
   4. Active malignancy or prior malignancy that was treated with chemotherapy
   5. History of a primary immunodeficiency disorder
   6. History of autoimmune cytopenias (i.e., ITP, AIHA)
   7. Coexisting medical condition that would place the child at increased risk for complications of study procedures
   8. Concurrent genetic or acquired disease or comorbidity(ies) that could require a future stem cell transplant
   9. Significant sensory (e.g., blindness, deafness, uncorrected hearing impairment) or motor (e.g., cerebral palsy) impairment
   10. Impaired renal or liver function as determined by serum creatinine >1.5mg/dL or total bilirubin >1.3mg/dL, except in patients with known Gilbert's disease
   11. Significant hematologic abnormalities defined as: Hemoglobin <10.0 g/dL, WBC < 3,000 cells/mL, ALC <1000/uL, Platelets <150 x 10e9/uL
   12. Known clinically relevant physical dysmorphology associated with neurodevelopmental conditions.
5. Current/Prior Therapy:

   a. History of prior cell therapy b. Current or prior use of IVIG or other anti-inflammatory medications with the exception of NSAIDs c. Current or prior immunosuppressive therapy i. No systemic steroid therapy that has lasted >2 weeks, and no systemic steroids within 3 months prior to enrollment. Topical and inhaled steroids are permitted.

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke Health; Geraldine Dawson, PhD, Principal Investigator — Duke Health; Jessica Sun, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | hCT-MSC Infusion
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: months] | 39.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 4
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 0
  Race: White | 7
  Race: More than one race | 0
  Race: Other | 1
  Race: Unknown or not reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Total Number of Infusion Reactions
Time Frame: 1 year
Measure: Number; unit: infusion reactions
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
infusion reactions | 1

2. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Severity of Infusion Reactions
Description: CTCAE is used to measure severity: 1= Mild, 2 = Moderate, 3 = Severe, 4 = Life-threatening, 5 = Death.
Time Frame: 1 year
Population: One participant experienced an infusion reaction.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 1
units on a scale | 1 (0)

3. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Total Number of Product-related Infections
Time Frame: 1 year
Measure: Number; unit: product-related infections
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
product-related infections | 0

4. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Severity of Product-related Infections
Description: CTCAE is used to measure severity: 1= Mild, 2 = Moderate, 3 = Severe, 4 = Life-threatening, 5 = Death.
Time Frame: 1 year
Population: No participants experienced a product-related infection.
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 0

5. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Number of Participants With Evidence of Alloimmunization Via Anti-HLA Antibodies
Time Frame: 1 year
Population: Three participants were not evaluable due to high levels of pre-existing HLA antibodies and one participant did not have post-infusion data collected.
Measure: Count of Participants; unit: Participants
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 9
Participants | 2

6. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Total Number of Graft vs. Host Disease (GVHD) Instances
Time Frame: 1 year
Measure: Number; unit: instances of GVHD
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
instances of GVHD | 0

7. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Severity of Graft vs. Host Disease (GVHD)
Description: CTCAE is used to measure severity: 1= Mild, 2 = Moderate, 3 = Severe, 4 = Life-threatening, 5 = Death.
Time Frame: 1 year
Population: No participants experienced GVHD.
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 0

8. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Total Number of Unexpected Adverse Events
Time Frame: 1 year
Measure: Number; unit: unexpected adverse events
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
unexpected adverse events | 0

9. Primary Outcome: Safety of hCT-MSC Infusion as Measured by Severity of Unexpected Adverse Events
Description: CTCAE is used to measure severity: 1= Mild, 2 = Moderate, 3 = Severe, 4 = Life-threatening, 5 = Death.
Time Frame: 1 year
Population: No participants experienced an unexpected adverse event.
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 0

10. Primary Outcome: Change in Pervasive Developmental Disorder Behavior Inventory Autism Composite Score (PDDBI)
Description: 6-month T score minus Baseline T score. PDDBI is designed to assess problem behaviors and social, language, and learning or memory skills of children who have been diagnosed with autism spectrum disorder. Raw scores are converted to T scores with a mean of 50 and standard deviation of 10, with a possible range of 10-100. Higher scores represent more severe problem behaviors. Therefore, a negative change in score indicates improvement.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: T score
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
T score | -5.00 [-9.92 to -0.08]

11. Primary Outcome: Change in VABS-3 (Vineland Adaptive Behavior Scales) Socialization and Communication Composite Score
Description: The change in the average of the Communication and Socialization Standard Subscale Scores on the Vineland Adaptive Behavior Scales (VABS-3) from the Comprehensive Interview form from baseline to six months. Higher scores indicate greater communication and/or socialization, with a range of 20 to 160 (mean = 100). A positive change in the scores indicates an improvement in communication and/or socialization.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
score on a scale | 3.83 [0.10 to 7.57]

12. Primary Outcome: Number of Participants Who Improved (Much Improved or Minimally Improved) on the Clinical Global Impression Scale (CGI)
Description: The number of participants who scored a 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the Clinical Global Impression Scale (CGI-I). The CGI-I score ranges from 1 to 7, where a lower score indicates greater improvement.
Time Frame: Baseline, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
Participants | 8

13. Primary Outcome: Change in Communicative Development Inventories (CDI-2)
Description: 6-month number of words produced minus baseline number of words produced. A positive change indicates improvement.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: words produced
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 12
words produced | 75.92 [16.10 to 135.73]

14. Primary Outcome: Change in Attention Abilities as Assessed Via Eye-tracking
Description: 6-month percentage of gaze directed towards social stimulus minus baseline percentage of gaze directed towards social stimulus. A negative change indicates improvement.
Time Frame: Baseline, 6 months
Population: Four participants did not have data available at both time points.
Measure: Mean (95% Confidence Interval); unit: percentage of gaze
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 8
percentage of gaze | -0.03 [-0.12 to 0.15]

15. Primary Outcome: Change in Brain Activity as Measured by EEG
Time Frame: Baseline, 6 months
Population: Data not collected.
Arm/Group | hCT-MSC Infusion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | hCT-MSC Infusion
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | hCT-MSC Infusion (N=12)
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Allergic reaction (Immune system disorders) | 1
Dental caries (Gastrointestinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 3
Food Aversions (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hyperactivity (Psychiatric disorders) | 1
Increased Aggression (Psychiatric disorders) | 1
Increased Hyperactivity (Psychiatric disorders) | 1
Increased Meltdowns (General disorders) | 1
Increased Repetitive Language (Psychiatric disorders) | 1
Increased Sensory Seeking Behaviors (Psychiatric disorders) | 1
Infections and Infestations (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Infusion related reaction (General disorders) | 1
Meltdowns (General disorders) | 1
Noncompliance (General disorders) | 1
Otitis media (Ear and labyrinth disorders) | 2
Repetitive Behaviors (Psychiatric disorders) | 2
Repetitive Language (Psychiatric disorders) | 1
Ritualistic Behaviors (Psychiatric disorders) | 2
Sensory Seeking Behaviors (Psychiatric disorders) | 2
Skin infection (Skin and subcutaneous tissue disorders) | 1
Sleep Difficulty (Nervous system disorders) | 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 8
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT04294290/Prot_SAP_000.pdf